CLINICAL TRIAL: NCT04090892
Title: Effects of Selective Percutaneous Muscle Lengthening on Gait in Children With Spasticity
Brief Title: Effects of Soft Tissue Lengthening on Gait in Children With Spasticity
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Susan Simpkins, Associate Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU 042014-068
Record Dates: First submitted 2014-08-06; First posted 2019-09-16 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-02

CONDITIONS: Muscle Spasticity
MeSH Terms: conditions — Muscle Spasticity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Persons with spasticity 4.0-20.11 years: Study personnel are not carrying out the surgical intervention but are assessing the outcomes of the surgery on gait and motor function.
  Interventions: Procedure: selective percutaneous muscle release

INTERVENTIONS:
Procedure: selective percutaneous muscle release — Children will be evaluated before and two times after they undergo a selective percutaneous myofascial release. Investigators make no determination about the need for the surgery or which muscles are released, nor do they participate in the surgery. The investigators are assess outcomes on gait and motor function.

SUMMARY:
This research project is being conducted to investigate changes in secondary impairments, functional mobility skills, and gait variables in children with spasticity following selective percutaneous myofascial lengthening. The research project proposed here will be the first to use instrumented three-dimensional motion analysis to investigate the effects of selective percutaneous myofascial lengthening on gait kinematics and kinetics. The objectives of the study are to:

1. Compare gait kinematics and kinetics in children and young adults with lower extremity spasticity before and after selective percutaneous myofascial lengthening to determine the effects of this procedure on functional mobility.
2. Identify changes in impairments and activity limitations following selective percutaneous myofascial lengthening .
3. Identify changes in a family or caregivers perceived quality of life after their child's selective percutaneous myofascial lengthening .

The aim of this study is to identify and describe the specific changes in secondary musculoskeletal impairments, activity limitations, and gait kinematics and kinetics after a selective percutaneous myofascial lengthening procedure. Gait kinematics and kinetics includes the motion of joints and body segments, and force and power, at each lower extremity joint, respectively. The results of this study will provide preliminary information on how this form of soft tissue lengthening affects functional mobility skills in children with spasticity. The study is expected to run for two years and the primary study endpoint is when participants have completed their second post- operative data collection session.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for an selective percutaneous myofascial lengthening procedure,
* Between the ages of 4.0 and 20.11 years old,
* Lower extremity spasticity,
* Able to ambulate 50 feet without a rest, with or without an assistive device, and with or without ankle foot orthoses (AFOs) and
* Able to follow one step directions.

Exclusion Criteria:

* Botox injections into any lower extremity muscle within three months of the scheduled selective percutaneous myofascial lengthening procedure,
* Lower extremity orthopedic surgery within 6 months of the scheduled selective percutaneous myofascial lengthening procedure,
* Visual impairment that interferes with maintaining a straight path while ambulating,
* Uncontrolled seizure disorder
* A change in medication that affects spasticity or ability to follow one step directions within three months of the scheduled selective percutaneous myofascial lengthening procedure.

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children between the ages of 4.0 and 20.11 years
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2016-05-10 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Kinematic Change is being assessed | Outcomes measures will be administered 4 weeks before surgery as a baseline
  Lower extremity joint angles at baseline before
Kinematic Change is being assessed | Outcomes measures will be administered then at 6 weeks after surgery to assess short term change
  Lower extremity joint angles after surgery
Kinematic Change is being assessed | Outcomes measures will be administered 6 months after surgery to assess long term change.
  Lower extremity joint angles after surgery

SECONDARY OUTCOMES:
Gross Motor Function Measure - Change is being assessed | Outcomes measures will be administered 4 weeks before surgery as a baseline
  Measures level of gross motor ability
Gross Motor Function Measure - Change is being assessed | Outcomes measures will be administered at 6 weeks after surgery to assess short term change
  Measures level of gross motor ability
Gross Motor Function Measure - Change is being assessed | Outcomes measures will be administered at 6 months after surgery to assess long term change.
  Measures level of gross motor ability

CONTACTS AND LOCATIONS:
Overall Officials: Susan D Simpkins, EdD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Children's Medical Center, Dallas, Texas, United States